CLINICAL TRIAL: NCT02663427
Title: Serological Screening of Gastric Cancer in Wuxi Region
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wuxi People's Hospital (Other)
Collaborators: Jiangsu Institute of Nuclear Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Z201501
Record Dates: First submitted 2016-01-17; First posted 2016-01-26 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Stomach Neoplasms
Keywords: pepsinogen Ⅰ; pepsinogen Ⅱ; gastric cancer screening; helicobacter pylori; gastrin
MeSH Terms: conditions — Stomach Neoplasms | interventions — Gastroscopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PG(-) and Hp(-) Group (Experimental): PG negative （pepsinogen（PG）Ⅰ > 70ng/ml or PGⅠ/PGⅡ >7.0）and Hp (helicobacter pylori) negative. A questionnaire survey are accomplished in 40-70 years old candidates. Eligible subjects are detected PG I and II, Hp-IgG antibody through serological examination. Gastroscope also accomplished in all participants.
  Interventions: Device: serological examination and gastroscope
- PG(-) and Hp(+) Group (Experimental): PG negative and Hp positive. A questionnaire survey are accomplished in 40-70 years old candidates. Eligible subjects are detected PG I and II, Hp-IgG antibody through serological examination. Gastroscope also accomplished in all participants.
  Interventions: Device: serological examination and gastroscope
- PG(+) and Hp(-) Group (Experimental): PG positive (PGⅠ ≤ 70ng/ml and PGⅠ/PGⅡ≤7.0) and Hp negative. A questionnaire survey are accomplished in 40-70 years old candidates. Eligible subjects are detected PG I and II, Hp-IgG antibody through serological examination. Gastroscope also accomplished in all participants.
  Interventions: Device: serological examination and gastroscope
- PG(+) and Hp(+) Group (Experimental): PG positive and Hp positive. A questionnaire survey are accomplished in 40-70 years old candidates. Eligible subjects are detected PG I and II, Hp-IgG antibody through serological examination. Gastroscope also accomplished in all participants.
  Interventions: Device: serological examination and gastroscope

INTERVENTIONS:
Device: serological examination and gastroscope

SUMMARY:
The purpose of this study is to determine whether detection of pepsinogen Ⅰand Ⅱ combined with Helicobacter pylori antibody, so-called ABC method , is fit on gastric cancer screening in community of Wuxi City.

DETAILED DESCRIPTION:
Gastric cancer is the third largest cause of cancer related deaths in China with about 350 ,000 gastric cancer-related deaths by gastric cancer in 2012. The studies from Japan and Korea have found gastric cancer screening, especially of the mass population, reduces mortality from gastric cancer, but the data is seldom in China. The ways include radiographic and endoscopic screening, although those methods were shown to reduce gastric cancer mortality, and was recommended as gold standard for population-based screening by Japan and Korea, but many problems have been pointed out: A serious drawback is low uptake of the target population; fear for radiation exposure(0.6 mSv), swallowing unpleasantness due to the use of barium meal, accidental fall during the examination and constipation, causing rare but more serious complications such as intestinal obstruction or diverticulitis after examination may account for the reasons for this low uptake, endoscopic screening is labor-intensive, more costly per examination as complete disinfection of the scope is mandatory, and requires a large number of well-trained experienced endoscopists.

Serological method, so-called ABC method , has been useful as gastric cancer preliminary screening in some areas, such as China, Japan and Korea. The major reasons are attributed to its simplicity, safety (radiation-free, discomfort free), and cost-efficiency. The ABC method is a blood test to stratify the risk of gastric cancer using the combination of H. pylori antibody and pepsinogen I and II, that was documented by large-scale studies in Japan. But the data was short in China, especially in the community.

ELIGIBILITY:
Inclusion Criteria:

Age 40-70 years old, men and women are not limited, and there are one of the following:

1. Hp infected.
2. Previously suffering from chronic atrophic gastritis, gastric ulcer, gastric polyps, hypertrophic gastritis, pernicious anemia and other precancerous diseases of the stomach.
3. First degree relatives of patients with gastric cancer.
4. Other risk factors for gastric cancer. (high salt, salted diet, smoking, heavy drinking, etc.)

Exclusion Criteria:

1. Severe heart, liver, kidney, dysfunction or mental disorders
2. History of gastric surgery (including surgery, minimally invasive EMR, ESD)
3. Use of PPI, acid preparation, stomach protecting agent in the first two weeks
4. The researchers considered inappropriate participants.
5. Informed consent cannot be attained

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
detection rate of gastric cancer among all group | through study completion, an average of 1 year

IPD SHARING:
Plan to Share IPD: Yes